CLINICAL TRIAL: NCT04118036
Title: A Phase 2 Study of Abemaciclib and Pembrolizumab in Recurrent Glioblastoma
Brief Title: Abemaciclib + Pembrolizumab In Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: safety concerns
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Patrick Wen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-351
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma
Keywords: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Surgery Arm (Experimental): In the surgical arm participants who require reoperation and have evidence of CDKN2A/B or C loss and intact RB from a prior tumor sample will receive
  * Pembrolizumab-prior to surgery, at predetermined dose and time point
  * Abemaciclib: every 12 hours from the day of pembrolizumab infusion to the morning of surgery
  * Post surgery Participants with receive
    * Abemaciclib, twice daily oral at specified dose for 21 day cycle
    * Pembrolizumab intravenous once in 21 day cycle (3 weeks)
  Interventions: Drug: Pembrolizumab; Drug: Abemaciclib
- Non Surgery Arm (Experimental): The treatment arm will be comprised of participants not requiring surgery.
  - Participants will receive treatment with
  * Abemaciclib, twice daily oral at specified dose for 21 day cycle
  * Pembrolizumab intravenous once in 21 day cycle (3 weeks)
  Interventions: Drug: Pembrolizumab; Drug: Abemaciclib

INTERVENTIONS:
Drug: Pembrolizumab — intravenously over 30 minutes every 21 days (+/- 3 days)
  Other Names: Keytruda
Drug: Abemaciclib — Oral 2 times a day
  Other Names: Verzenio

SUMMARY:
This research study is studying a combination therapy as a possible treatment for recurrent glioblastoma (GBM), a brain tumor that is growing or progressing despite earlier treatment.

This study will involve participants with recurrent glioblastoma at their first relapse enrolled in two arms including patients who require reoperation and patients not requiring surgery.

This research study involves a combination of two drugs:

* Pembrolizumab (MK3475)
* Abemaciclib (LY2835219)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease.

"Investigational" means that the drug is being studied.

Many brain cancers show over expression of a protein called cyclin D1. That means that the body makes too much cyclin D1, which affects enzymes called CDK 4 and CDK 6. Enzymes are substances in the body that help reactions between cells happen. Too much cyclin D1 triggers CDK 4 and CDK 6 to make more cells than normal. This extra cell production leads to the growth of tumors.

In laboratory studies, abemaciclib was able to enter the brain, stop CDK 4 and CDK 6 from making cells, and slow growth of glioblastoma in mice.

Pembrolizumab (MK-3475) has been studied in lab experiments and in other types of cancer. Information from these studies suggests that Pembrolizumab (MK-3475) may be beneficial inrecurrent glioblastoma (GBM). Pembrolizumab (MK-3475) is a humanized monoclonal antibody. An antibody is a common type of protein made in the body in response to a foreign substance. Antibodies attack foreign substances and protect against infection. Antibodies can also be produced in the laboratory for use in treating patients; an antibody that is made in the lab is also known as a humanized monoclonal antibody that is designed to block the action of the receptor, PD-1. PD-1 works to help tumor cells continue to grow and multiply. There are now several approved antibodies for the therapy of cancer and other diseases.

.

ELIGIBILITY:
Inclusion Criteria:

* All participants must meet the following criteria on screening examination to be eligible to participate in the study:

  * Participants must be able to understand and willing to sign a written informed consent document.
  * Participants must be able to adhere to the dosing and visit schedules, and agree to record medication times accurately and consistently in a daily diary.
  * Participants must be at least 18 years old on day of signing informed consent.
  * Participants must have a Karnofsky Performance Status (KPS) ≥ 70 (see Appendix A).
  * Participants must be able to swallow oral medications.
* Nature of illness and treatment history

  * Participants must have histologically confirmed diagnosis of glioblastoma or variants. Participants will not be eligible if the prior diagnosis was low-grade glioma and a subsequent histological diagnosis of glioblastoma or variants was made (e.g. secondary GBM).
  * To be eligible for the study all participants (Cohort 1 and 2) are required to provide genomic profiling data from a sequencing-based assay and must include reporting of the RB1 gene in explicit terms within the report. Only sequencing assays that include coverage of all exons of the RB1 gene are able to be utilized (most commonly called a targeted exome assay; e.g. Oncopanel, Impact, FoundationOne). In addition, patients must provide a report of copy assessment which reports status of RB1. The reporting may be from a copy array (ideally Oncoscan SNP array or Agilent array CGH) or can also be from sequencing assay if copy status is explicitly provided with quantitative information regarding the status of relevant genes.
  * Inactivation of CDKN2A/B or C in the tumor by homozygous deletion (evidence for more than single copy loss for any of the genes defined as copy array log2 ratio of <0.3 by copy array; or from sequencing data with sufficient coverage for evaluation). Rearrangement/evidence or intragenic breaks by copy or sequencing assay also will be considered eligible for study (any copy status).
  * Validation of wild-type RB status (no deletion/losses more than single copy by copy number or sequencing data; and/or no inactivating mutations or rearrangement by sequencing).
  * Participants must be at first relapse of GBM. Relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy). The intent therefore is that patients had no more than 1 prior therapy (initial treatment). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered to constitute 1 relapse.
  * Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.

    * For Cohort 2 subjects, CT or MRI within 14 days prior to study registration. For Cohort 2, corticosteroid dose must be stable or decreasing for at least 5 days prior to the scan. If steroids are added or the steroid dose is increased between the date of the screening MRI or CT scan and the start of treatment, a new baseline MRI or CT is required.
    * For Cohort 1 subjects, CT or MRI should be performed ideally within 14 days prior to study registration, but because the screening MRI for this subset of subjects will not be used for evaluation of response, it is acceptable for this MRI/CT to have been performed greater than 14 days prior to registration if unavoidable. Furthermore, for this same reason, fluctuation in corticosteroid dose around this MRI does not warrant repeat scan so long as there is documented unequivocal evidence of tumor progression available.
  * Confirmation of availability of sufficient tissue from a prior surgery demonstrating glioblastoma or variants for correlative studies is required prior to enrollment; these samples must be sent to the DFCI Coordinating Center within 60 days of registration.

The following archived tissue is required for Cohort 2 patients:

--- 20 unstained formalin fixed paraffin embedded (FFPE) sections (standard 5 micrometer thickness).

The following amount of archived tissue is required for Cohort 1 patients:

* 20 unstained formalin fixed paraffin embedded (FFPE) sections (standard 5 micrometer thickness)
* For Cohort 1 subjects, there must be > 2cm2 enhancing tissue available for resection and submission for study correlatives as determined by local treating team. NOTE: if the above-mentioned tissue is not available from the most recent surgery revealing GBM, participants may be enrolled with tissue available from any prior surgery revealing GBM with prospective approval from the Overall PI. An interval of at least 12 weeks from the completion of radiation therapy to start of study drug unless there is a new area of enhancement consistent with recurrent tumor outside the radiation field (defined as the region outside the high-dose region or 80% isodose line) or there is unequivocal histologic confirmation of tumor progression.

  * Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
  * From the projected start of scheduled study treatment, the following time periods must have elapsed:
* 4 weeks or 5 half-lives (whichever is shorter) from any investigational agent;
* 4 weeks from cytotoxic therapy (except 23 days for temozolomide; 6 weeks from nitrosoureas);
* 4 weeks from antibodies;
* 4 weeks or 5 half-lives (whichever is shorter) from other anti-tumor therapies.
* 2 days from Novo-TTF

  * Participants with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of progressive disease based upon nuclear imaging, MR spectroscopy, perfusion imaging or histopathology.
  * Participants having undergone recent resection or open biopsy or stereotactic biopsy of recurrent or progressive tumor will be eligible for Cohort 2 as long as the following conditions apply:
* They have recovered from the effects of surgery.
* Residual disease following resection of recurrent tumor is not mandated for eligibility.

  * Clinical labs - performed within 14 days prior to registration
  * Hematology:

    * Leukocytes ≥ 3 K/µL
    * Absolute neutrophil count (ANC) ≥ 1.5 K/µL
    * Platelet count ≥ 100 K/µL
    * Absolute Lymphocyte Count ≥ 0.5 K/µL
    * Hemoglobin ≥ 8.0 g/dL
  * Biochemistry:

    * Total serum calcium (corrected for serum albumin as needed) or ionized calcium within institution's normal range, or correctable with supplements.
    * Magnesium within institution's normal range, or correctable with supplements.
    * AST (SGOT) and ALT (SGPT) ≤ 2.5 x institution's ULN (or ≤ 5 X institutional ULN for subjects with Gilberts syndrome)
    * Serum bilirubin ≤ 1.5 x institution's ULN
    * Serum creatinine ≤ 1.5 x institution's ULN or calculated 24-hour creatinine clearance ≥ 50 mL/min
    * Serum amylase ≤ 1.5 x institution's ULN
    * Serum lipase ≤ 1.5 x institution's ULN
    * Serum albumin ≥ 2.5 g/dL
  * Coagulation studies:

    * INR < 2.0
    * PTT ≤ institution's ULN, unless receiving therapeutic low molecular weight heparin or oral factor Xa inhibitors.
  * Other illnesses

    -- Patients with prior or concurrent malignancy whose natural history or treatment does not give the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  * Pregnancy and Reproduction

    * The effects of abemaciclib and pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) must agree to use a medically approved contraceptive method during the treatment period and for 120 days following the last dose of study drug. Men must agree to use a reliable method of birth control and to not donate sperm during the study and for at least 120 days following the last dose of study drug.
    * Women of child-bearing potential must have a negative serum pregnancy test within 7 days prior to first dose of abemaciclib.

Exclusion Criteria:

* Participants who meet any of the following criteria will not be eligible for admission into the study.
* Pathology

  * Prior evidence of 1p/19q co-deletion.
  * IDH1/2 mutation in any prior biopsy.
  * Tumor primarily localized to the brainstem or spinal cord.
  * Presence of diffuse leptomeningeal disease or extracranial disease.
* Previous therapies

  * Participants who have received prior treatment with a CDK4/6 inhibitor (e.g. abemaciclib, palbociclib).
  * Participants who have received anti-VEGF targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL184, sunitinib etc.).
  * Participants who have received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
  * Participants who have received prior interstitial brachytherapy, implanted chemotherapy, stereotactic radiosurgery or therapeutics delivered by local injection (including intra-tumoral vaccines) or convection enhanced delivery.
* Concomitant medications

  * Participants requiring treatment with high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 2 weeks of start of study drug.
  * Participants who have received systemic immunosuppressive treatments, aside from systemic corticosteroids (such as methotrexate, chloroquine, azathioprine, etc.) within six months of start of study drug.
  * Participants taking an enzyme-inducing anti-epileptic drug (EIAED): phenobarbital, phenytoin, fosphenytoin, primidone, carbamazepine, oxcarbazepine, eslicarbazepine, rufinamide, and felbamate. Participants must be off any EIAEDs for at least 14 days prior to starting study drug. A list of EIAEDs and other inducers of CYP3A4 can be found in Appendix D.
  * Participants taking a drug known to be a strong inhibitor or inducer of isoenzyme CYP3A (Appendix D). Participant must be off CYP3A inhibitors and inducers for at least 7 days prior to starting study drug. NOTE: participants must avoid consumption of Seville oranges (and juice), grapefruits or grapefruit juice, grapefruit hybrids, pummelos and exotic citrus fruits from 7 days prior to the first dose of study drug and during the entire study treatment period due to potential CYP3A4 interaction.
  * Participants receiving any other investigational agents.
  * Current use of herbal preparations/medications, including but not limited to: St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, ginseng. Participants should stop using these herbal medications 7 days prior to first dose of study drug.
  * Current use of warfarin sodium or any other coumadin-derivative anticoagulant. Participants must be off Coumadin-derivative anticoagulants for at least 7 days prior to starting study drug. Low molecular weight heparin and Factor Xa inhibitors are allowed.
* Other illnesses

  * History of allergic reactions attributed to compounds of similar chemical or biologic composition to abemaciclib and/or pembrolizumab.
  * History of intratumoral or peritumoral hemorrhage if deemed significant by the treating investigator. If there are questions, the treating investigator should contact the study Overall P.I., Patrick Wen, MD, at 617-632-2166.
  * Uncontrolled intercurrent illness.
  * Participant has an active infection requiring systemic therapy and/or known viral infection (for example, human immunodeficiency virus antibodies, hepatitis B surface antigen or hepatitis C antibodies).
  * Participant with a known history of active TB (Bacillus Tuberculosis).
  * Participant with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
  * Participant with a diagnosis of immunodeficiency, including a known history of Human Immunodeficiency Virus (HIV).
* Participants who have received a live vaccine within 30 days prior to start of study treatment.

  -- Participants with diarrhea ≥ CTCAE grade 2
* Participant has active cardiac disease including any of the following:

  * Angina pectoris that requires the use of anti-anginal medications.
  * Ventricular arrhythmias except for benign premature ventricular contractions.
  * Supraventricular and nodal arrythmias requiring a pacemaker or not controlled with medication.
  * Conduction abnormality requiring a pacemaker.
  * Valvular disease with document compromise in cardiac function.
  * Symptomatic pericarditis.
  * Participant has a history of cardiac dysfunction including any of the following:

    * Myocardial infarction within the last 6 months prior to start of study drug, documents by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function.
    * History of documents congestive heart failure (New York Heart Association functional classification III-IV, see Appendix I).
    * Documented cardiomyopathy.
    * Congenital long QT syndrome.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of abemaciclib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection). Participants with unresolved diarrhea ≥ CTCAE grade 2 will be excluded as previously indicated.

  * Participants who have undergone major systemic surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
  * Participants who are pregnant or breastfeeding.
  * Participants with history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug or gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of start of study drug.
  * Has known history of, or any evidence of, active non-infectious pneumonitis.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
TIL density in tumor tissue (surgery) | Day 1-Post Surgery
  One-sided Wilcoxon test
Progression Free Survival 6 months (non surgery) | 6 months
  Kaplan Meier curves
Radiographic response rate (non surgery) | 2 years
  RANO Criteria
Median progression free survival | 2 Years
Overall survival | From date of first dose (date of first post-surgery treatment for participants in Cohort 1) to date of death due to any causeup to 100 months
  calculated using standard statistical methods
Tumor cell death (Surgery) | 2 years
  Effects of abemaciclib and pembrolizumab on tumor cell proliferation and tumor cell death will be measured using immunohistochemistry for pRB1, Ki-67 and Cleaved Caspase 3
tumor cell proliferation (surgery) | 2 years
  Effects of abemaciclib and pembrolizumab on tumor cell proliferation and tumor cell death will be measured using immunohistochemistry for pRB1, Ki-67 and Cleaved Caspase 3

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu